CLINICAL TRIAL: NCT03432299
Title: Radiofrequency Ablation of Low Risk Papillary Thyroid Microcarcinoma: Safety and Efficacy
Brief Title: Radiofrequency Ablation of Low Risk Papillary Thyroid Microcarcinoma
Acronym: RFAforPTMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-hoon Kim, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-RFA-PTMC
Record Dates: First submitted 2018-01-22; First posted 2018-02-14 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Papillary Thyroid Microcarcinoma; Thyroid Cancer
Keywords: Thyroid Diseases; Radiofrequency Ablation
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma; Thyroid Neoplasms; Thyroid Diseases | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFA for PTMC (Experimental): Group who will undergo RFA after diagnosis of PTC
  Interventions: Procedure: RFA for PTMC

INTERVENTIONS:
Procedure: RFA for PTMC — Radiofequency ablation for papillary thyroid microcarcinoma will be performed using the system including radiofrequency generator and internally cooled electrode.

SUMMARY:
This is a single center prospective clinical trial with regard to efficacy and safety of radiofrequency ablation of papillary thyroid microcarcinoma.

DETAILED DESCRIPTION:
For treatment of papillary thyroid microcarcinoma (PTMC), radiofrequency ablation (RFA) will be performed with the supine position and neck extended under ultrasonogrphic guidance. Before RFA, local anesthesia will be performed. RFA system including radiofrequency generator (VIVA RF system, STARmed, Goyang-si, Korea) and internally cooled electrode (star RF electrode, STARmed, Goyang-si, Korea) will be used. With regard to RFA procedure, moving shot technique and hydrodissection, if indicated, will be used. After RFA, follow-up will be performed using ultrasonography, serum thyroid function test, and questionnaire for quality of life by face-to-face interview at 2 months, 6, 12, 18, 24 months during the first 2 years after RFA, and yearly afterwards.

ELIGIBILITY:
Inclusion Criteria:

* who agrees to the consent form
* aged from 19 to 60 years old
* who has been diagnosed with Bethesda category V or VI by fine needle aspiration or needle biopsy
* whose thyroid cancer is 1 cm or smaller than 1 cm length
* who does not have lymph node or distant metastasis
* whose thyroid cancer does not have extrathyroidal extension
* in whom it seems technically possible to completely ablate thyroid cancer using RF

Exclusion Criteria:

* who cannot routinely followed up according to the study schedule
* who has been with Bethesda category I, II, III, or IV by fine needle aspiration or needle biopsy.
* who has hyperthyroidism that requires treatment
* who has bleeding tendency
* multifocal papillary thyroid microcarcinoma
* who is pregnant

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of tumor size | baseline, 2, 6, 12, 18, 24 months during the first two years after RFA, and yearly afterwards upto 10 years
  Maximal dimension (mm) of ablation zone on Ultrasonography

SECONDARY OUTCOMES:
Development of Metastasis | baseline, 2, 6, 12, 18, 24 months during the first two years after RFA, and yearly afterwards upto 10 years
  Cervical Lymph node metastasis on Ultrasonography or other distant metastasis
Change of Quality of Life | baseline, 2, 6, 12, 18, 24 months during the first two years after RFA, and yearly afterwards upto 10 years
  Score on a Korean version of a thyroid-specific Quality-of-life Questionnaire Scale in Thyroid Cancer Patients
Incidence of potential side effects from RFA | baseline, 2, 6, 12, 18, 24 months during the first two years after RFA, and yearly afterwards upto 10 years
  rate of patients who underwent potential side effects from RFA

CONTACTS AND LOCATIONS:
Overall Officials: Ji-hoon Kim, MD,Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JY, Na DG, Sim JS, Sung JY, Cho SW, Park DJ, Park YJ, Kim JH. A Prospective Clinical Trial of Radiofrequency Ablation in Patients with Low-Risk Unifocal Papillary Thyroid Microcarcinoma Favoring Active Surveillance Over Surgery. Thyroid. 2024 Sep;34(9):1126-1136. doi: 10.1089/thy.2024.0098. PMID 39212950